CLINICAL TRIAL: NCT01157767
Title: A Feasibility Study of the Effects of a Directed Exercise Program of Breast Cancer Patients Undergoing Chemotherapy With or Without Radiation
Brief Title: Exercise Program of Breast Cancer Patients Undergoing Chemotherapy With or Without Radiation
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 10-062
Record Dates: First submitted 2010-07-06; First posted 2010-07-07 (Estimated); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer
Keywords: exercise; lymphedema; post-operative chemotherapy; post-operative radiation; 10-062
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- breast pts who have undergone surgery: This will be a feasibility study designed to evaluate the compliance of an at-home, directed exercise program and its influence on physical measures during post-operative adjuvant chemotherapy and radiation (if applicable).
  Interventions: Other: standardized regimen of exercises, including a warm-up period, ROM arm exercises, and strength training exercises.

INTERVENTIONS:
Other: standardized regimen of exercises, including a warm-up period, ROM arm exercises, and strength training exercises. — Module I is a group of arm movements. It consists of stretching exercises coordinated with breathing exercises to restore their physical mobility, range of motion and flexibility of shoulders. Module I is to be performed daily. In Module II the exercises are a series of copyrighted, sequential movements designed to put the body in proper alignment. It is a special series of muscle movements to help establish better body alignment, as well as increased strength and flexibility of one's arms, legs, and spine, each exercise is 4 repetitions. Module III is the walking and the resistance weight training program. The walking program is whole body exercise, multi-joint, weight-bearing, low impact and for beginners to advanced.

SUMMARY:
The purpose of this study is to study if a patients follows an exercise program specifically designed for them during the time of their treatment after surgery. Their ability to follow the program and its influence on their weight maintenance and early post-operative lymphedema rates will also be studied. Lymphedema is a condition in which excess fluid collects in tissue and causes swelling of the arm(s).

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible if they have any of the following surgical procedures performed by an attending on the Breast Service:

SLNB alone Axillary lymph node dissection (ALND) alone Total Mastectomy TM (+/- reconstruction) with SLNB or ALND Breast conserving therapy (BCT) with SLNB or ALND

* Age > 18 years
* Planned to undergo adjuvant post-operative chemotherapy with or without radiation at MSKCC and have not yet started chemotherapy

Exclusion Criteria:

* Undergoing TM or BCT without SLNB
* Having had prior breast cancer treated with surgery
* Unable to participate in a exercise program related to other medical problems
* More than 8 weeks post surgery.
* Having a concurrent cancer in addition to breast cancer
* Who have had any type of chemotherapy in the past two years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects may be identified in advance by a member of the patient's treatment team, the principal investigator, or research team at Memorial Sloan-Kettering Cancer Center (MSKCC).
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2010-05-11 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-08-23 (Actual)

PRIMARY OUTCOMES:
To evaluate compliance with and demonstrate the feasibility of an at-home, directed exercise program during adjuvant chemotherapy and radiation (if applicable). | 2 years

SECONDARY OUTCOMES:
To describe how this exercise program affects weight maintenance and percent body fat during adjuvant chemotherapy and radiation. | 2 years
To describe how this exercise program affects early post-operative lymphedema rates, monitoring the strength training specifics -including the number of repetitions and sets of each exercise, frequency, and order of exercises. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Heerdt, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm